CLINICAL TRIAL: NCT05988593
Title: Testing the Cognitive Facilitation Effect by Dietary Supplementation of MelaGene+ Drink
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CMUH111-REC3-127
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Cognitive Change

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo drink (Placebo Comparator)
  Interventions: Dietary Supplement: placebo
- MelaGene+ (Experimental)
  Interventions: Dietary Supplement: MelaGene+

INTERVENTIONS:
Dietary Supplement: placebo — consume one bottle (30 mL) per day
  Arms: placebo drink
Dietary Supplement: MelaGene+ — consume one bottle (30 mL) per day
  Other Names: Melaleuca-MelaGene+
  Arms: MelaGene+

SUMMARY:
To assess the efficacy of MelaGene+ on cognitive performance

ELIGIBILITY:
Inclusion Criteria:

* 20 to 65-year-old males or females

Exclusion Criteria:

* Participants are breastfeeding, pregnant or planning to become pregnant during the test (self-report)
* Participants with heart, liver, kidney, endocrine and other major organic diseases (self-reported)
* Participants take drugs for a long time (self-report)
* Participants with mental illness or have undergone brain surgery
* Participants still can not clearly see words with 12pt on computer after corrected vision

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
The change of Match to sample test | Change from Baseline match to sample test value at 8 weeks
  The number of memorized cards was utilized to measure Match to sample test value.
The change of Trail making test | Change from Baseline Trail making test value at 8 weeks
  The time of finishing actions was utilized to measure Trail making test value.
The change of Processing speed test | Change from Baseline Processing speed test value at 8 weeks
  The number of pressing buttons was utilized to measure Processing speed test value.
The change of Mnemonic Similarity Task | Change from Baseline Mnemonic Similarity Task value at 8 weeks
  The proportion of correction about ability on memorizing old things was utilized to measure Mnemonic Similarity Task value.
The change of facial expression cuing task | Change from Baseline facial expression cuing task value at 8 weeks
  The correction of evaluation on facial emotion was utilized to measure facial expression cuing task value.
The change of State-trait anxiety inventory | Change from Baseline State-trait anxiety inventory value at 8 weeks
  The scores of anxiety state was utilized to measure State-trait anxiety inventory value.
The change of score of fatigue | Change from Baseline PSS (The Perceived Stress Scale)-14 value at 8 weeks
  The PSS (The Perceived Stress Scale)-14 questionnaire was utilized to measure fatigue condition.
The change of score of life quality | Change from Baseline WHOQOL-BREF (The World Health Organization Quality of Life Brief Version) value at 8 weeks
  The WHOQOL-BREF (The World Health Organization Quality of Life Brief Version) questionnaire was utilized to measure life quality.

CONTACTS AND LOCATIONS:
Overall Officials: Jing-Ling Li, Principal Investigator — China Medical University, China
Locations (1):
- China Medical University, Taichung, Taiwan